CLINICAL TRIAL: NCT06105385
Title: Investigation of the Instant Effects of the Suboccipital Myofascial Release Technique on Cervical Proprioception, Joint Range of Motion and Balance in Young Adults
Brief Title: Suboccipital Myofascial Release Technique in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fatih Tekin, Assist. Prof., Pamukkale University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Myofascial Release
Record Dates: First submitted 2023-10-16; First posted 2023-10-27 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Myofascial Release
Keywords: Suboccipital Myofascia; Release Technique; Cervical Proprioception; Range of Motion; Balance

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First (Experimental): Suboccipital Myofascial Release Technique will be applied to this group first. After the intervention in this group is completed, the transition to the other crossover group will be made.
  Interventions: Other: Suboccipital Myofascial Release Technique
- Second (Experimental): Once the intervention to the first group is completed, the second intervention "Suboccipital Myofascial Release Technique" will be applied to this group.
  Interventions: Other: Suboccipital Myofascial Release Technique

INTERVENTIONS:
Other: Suboccipital Myofascial Release Technique — With the patient in a supine position, the therapist sits behind the patient with his or her forearms on the treatment table. The therapist places his fingers between the occiput and axis, with his fingers in semi-flexion (2nd, 3rd and 4th fingers), and continues to hold his hands on the occiput until relaxation is achieved in the suboccipital muscles. A light traction is applied at the end of the technique. Average application time is 4-5 minutes.

SUMMARY:
When the literature is examined, although it is known that the suboccipital muscles are rich in proprioceptive receptors and have significant effects on balance, the effects of myofascial and neural relaxation of the suboccipital muscles on balance and proprioception are not fully understood. In this study, the investigators aim to examine the immediate effects of the SMV technique on balance and proprioception in young adults. With this study, by revealing the effects of the SMV technique on balance and proprioception, a different treatment option will be offered to clinicians working in the field of physical therapy and rehabilitation and interested in the rehabilitation of patients who may have balance and proprioception problems. It will also provide insight to academics working in this field in terms of the applicability of this technique among different patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Being healthy and not having one of the diseases specified in the exclusion criteria

Exclusion Criteria:

* Individuals with neck pain, neck trauma (fracture, whiplash syndrome), balance and proprioception problems, vestibular system problems, vertigo, cervical surgery, vision and hearing problems, any rheumatological, orthopedic, cardiovascular and neurological problems that may affect the cervical region

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2023-10-12 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-12 (Actual)

PRIMARY OUTCOMES:
Joint Position Error Measurement | Before and Immediately After the Treatment Process
  The Cervical Joint Position Error Test is a measurement tool used to clinically assess an individual's cervicocephalic proprioception ability. Cervicocephalic proprioception describes one's sense of position of their head and neck in space.
Cervical Joint Range of Motion Measurement | Before and Immediately After the Treatment Process
  Cervical joint movement, cervical flexion, extension, right and left rotation, right-left lateral flexion movement will be measured with the help of a suitable goniometer.
Balance Assessment | Before and Immediately After the Treatment Process
  Portable computerized kinesthetic balance device (SportKAT) examines balance in 2 main parameters: static and dynamic, and 4 main parameters: forward-backward, right-left. SporKAT consists of a platform on the ground and a screen designed to be directly in front of the patient, 1 meter away from the patient. After the pressure values of the platform are adjusted, the content of the test is explained to the patient and the patient is placed on the platform with bare feet, and then the patient's feet are adjusted to the specified places on the platform. During the test, the patient is asked to try to keep the x (cross) sign on the screen in the middle of the circle visible on the screen for 30 seconds. The test is terminated after 30 seconds. Higher balance scores indicate that the person's balance is more impaired.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Tekin, Ass. Prof., Study Chair — Faculty Member
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)